CLINICAL TRIAL: NCT01854567
Title: A 1-Year, Multicenter, Randomized, Open-Label Controlled Study to Evaluate the Efficacy and Safety of Cord Blood Cells Expanded With MPCs for Hematopoetic Recovery in Patients With Hematologic Malignancies After Myeloablative Treatment
Brief Title: P3 Study of Umbilical Cord Blood Cells Expanded With MPCs for Transplantation in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB-AB006; 2012-0166 (Other: UT MDACC)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; Hodgkin's Disease
Keywords: Cord Blood; Stem Cells; MPC; Mesoblast; Expanded; AML; ALL; NHL; Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Infusion of one MPC expanded cord unit and one unexpanded cord unit.
  Interventions: Biological: Infusion of one MPC expanded cord unit and one unexpanded cord unit
- Control (Active Comparator): Infusion of two unexpanded cord blood units.
  Interventions: Biological: Infusion of two unexpanded cord blood units.

INTERVENTIONS:
Biological: Infusion of one MPC expanded cord unit and one unexpanded cord unit — Infusion of one MPC expanded cord unit and one unexpanded cord unit.
  Arms: Active
Biological: Infusion of two unexpanded cord blood units. — Umbilical Cord Blood.
  Arms: Control

SUMMARY:
The study investigates the time to engraftment of a mesenchymal expanded cord blood unit in patients with hematologic malignancies undergoing transplantation with myeloablative conditioning.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have one of the following:

  * Acute myelogenous leukemia (AML) in complete morphological remission at study screening (Complete Remission with Incomplete Platelet Recovery (CRp) acceptable).
  * Acute lymphoblastic leukemia (ALL) in complete morphological remission at study screening (Complete Remission with Incomplete Platelet Recovery (CRp) acceptable).
  * Non-Hodgkin's lymphoma (NHL): High risk subjects with responsive disease after first relapse. High risk includes those with Burkitt's Lymphoma and those with extensive marrow involvement at diagnosis-precluding autologous transplant.
  * Hodgkin's disease: High risk subjects with responsive disease after first relapse.
* Minimum Karnofsky Scale
* Subject must weigh at least 20 kg
* Up to 65 years of age
* Adequate major organ system function

Exclusion Criteria:

* Pregnancy and/or lactating
* Suitable, 6/6 HLA matched related sibling donor available
* Previous participation in a stem cell study within last 30 days

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Time to Neutrophil and Platelet Engraftment | 100 days

SECONDARY OUTCOMES:
Proportion of subjects with neutrophil recovery at day 26, platelet recovery at day 60 and subjects alive at day 100 | 100 days
Percentage of patients with primary graft failure | 100 days

OTHER OUTCOMES:
Incidence and severity of acute Graft Versus Host Disease | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Donna Skerrett, MD, MS, Study Director — Mesoblast, Ltd.; Elizabeth J. Shpall, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - University of Miami Health System Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell-New York Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Case Western, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Center at Methodist Healthcare System, San Antonio, Texas